CLINICAL TRIAL: NCT05306379
Title: A Single Center, Open Label, Phase 1 Drug-Drug Interaction Study to Investigate the Effects of Voclosporin on the Pharmacokinetics of Simvastatin in Healthy Volunteers
Brief Title: Drug-Drug Interaction Study to Investigate Effects of Voclosporin on Pharmacokinetics of Simvastatin
Acronym: Statin-DDI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aurinia Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AUR-VCS-2021-02
Record Dates: First submitted 2022-02-07; First posted 2022-04-01 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Drug-drug Interaction
Keywords: voclosporin; simvastatin; pharmacokinetics; drug effects; drug interactions
MeSH Terms: interventions — Simvastatin; voclosporin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Voclosporin/Simvastatin (Experimental): Subjects will receive a single oral dose of 40 mg simvastatin (given as two 20 mg tablets) in the morning of Day 1 and Day 8.
  Subjects will receive voclosporin administered as an oral 23.7 mg dose (three 7.9 mg capsules) twice-daily for 7 days from the morning of Day 2 until the evening of Day 8.
  Interventions: Drug: Simvastatin; Drug: Voclosporin

INTERVENTIONS:
Drug: Simvastatin — Oral dose 40 mg
Drug: Voclosporin — Oral dose 23.7 mg twice daily

SUMMARY:
A single-center, open-label, Phase 1, drug-drug interaction study to investigate the effect of voclosporin on the pharmacokinetics of simvastatin and simvastatin acid in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Healthy male or female subjects aged >=18 and <=55 years
* Body mass index >=18.0 and <32 kg/m2

Exclusion Criteria:

* Abnormal ECG and/or prolonged QT interval
* Subjects using nicotine products within 3 months prior to screening
* Subjects who have lost or donated >450 mL of whole blood or blood products within 30 days prior to the Screening Visit.
* Use of any prescription medication within 14 days prior to the first dose of study medication, or any over-the-counter products (including natural health products, e.g., food supplements, vitamins, herbal supplements) within 7 days prior to the first dose of study medication, except for topical products without significant systemic absorption.
* Use of any drugs or substances known to induce or inhibit hepatic drug metabolism within 28 days prior to administration of the study medication
* Consumption of grapefruit or grapefruit juice, pomelo or star fruit within 7 days of first dose of study drug on Day 1
* Use of hormonal contraception or hormone replacement therapy within 14 days prior to first dose of study drug.
* No COVID-19 vaccines are allowed within 28 days prior to first dose of study drug.
* History of or current alcohol abuse or drug addiction
* Subjects who are pregnant or breast feeding
* Subjects who have received any investigational drug within 30 days or 5 half-lives of the drug (whichever is longer) prior to screening.
* Subjects who have any significant health issues as deemed by their treating physician/investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2022-04-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of simvastatin and simvastatin acid (Cmax) | 9 days
  To evaluate the potential effect of multiple oral doses of voclosporin on the single-dose PK of simvastatin and the active metabolite simvastatin acid. Maximum observed concentration (Cmax).
Pharmacokinetics of simvastatin and simvastatin acid (AUC) | 9 days
  To evaluate the potential effect of multiple oral doses of voclosporin on the single-dose PK of simvastatin and the active metabolite simvastatin acid. Area under the concentration-time curve (AUC) from time zero to infinity.
Pharmacokinetics of simvastatin and simvastatin acid (AUC) | 9 days
  To evaluate the potential effect of multiple oral doses of voclosporin on the single-dose PK of simvastatin and the active metabolite simvastatin acid. Area under the concentration-time curve (AUC) time zero to last quantifiable concentration.

SECONDARY OUTCOMES:
Pharmacokinetics of voclosporin (Cmax) | 9 days
  To evaluate voclosporin blood concentrations - Cmax.
Pharmacokinetics of voclosporin (AUC) | 9 days
  To evaluate voclosporin blood concentrations - AUC from time zero to 12 hours.
Pharmacokinetics of voclosporin (Tmax) | 9 days
  To evaluate voclosporin blood concentrations - Time to reach maximum observed plasma concentration (Tmax).
Pharmacokinetics of voclosporin (Ctrough) | 9 days
  To evaluate voclosporin blood concentrations - Trough concentration (Ctrough) at the end of a dosing interval at steady state.
Pharmacokinetics of voclosporin (CL/F) | 9 days
  To evaluate voclosporin blood concentrations - apparent clearance (CL/F).
Number of participants with abnormal laboratory test results | Up to 2 weeks
  Number of subjects with abnormal laboratory test results (eg., hematology, biochemistry and urinalysis) will be assessed
Number of participants with abnormal vital signs | Up to 2 weeks
  Number of participants with abnormal vital signs (eg., blood pressure, heart rate, body temperature, respiratory rate) will be assessed
12-Lead Electrocardiogram Assessment | Up to 2 weeks
  Standard 12-lead electrocardiograms (eg., QTcF interval) will be summarized by observed value and change from baseline values.

CONTACTS AND LOCATIONS:
Overall Officials: Winnie Lim, Study Director — Aurinia Pharmaceuticals Inc.
Locations (1):
- Labcorp Clinical Research Unit, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No